CLINICAL TRIAL: NCT00896909
Title: Evaluation of HER2 Mutations in Patient Tumors From E2598
Brief Title: HER-2 Mutations in Tumor Samples From Patients With Advanced Non-Small Cell Lung Cancer Treated on Clinical Trial ECOG-2598
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000476582; ECOG-E2598T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gene Expression Profiling; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Collecting samples of tumor tissue from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at HER-2 mutations in tumor samples from patients with advanced non-small cell lung cancer being treated with trastuzumab on clinical trial ECOG-2598.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate clinical response to trastuzumab (Herceptin®) with the presence of mutation in the HER-2 kinase domain in tumor samples from patients with advanced non-small cell lung cancer treated on protocol ECOG-2598.
* Correlate mutations with time to progression and survival of these patients.

OUTLINE: This is a multicenter study.

Tissue specimens are analyzed by polymerase chain reaction to assess mutations in the HER-2 gene. Laboratory/biomarker analysis data is correlated with clinical data from protocol ECOG-2598.

PROJECTED ACCRUAL: A total of 22-44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer meeting ≥ 1 of the following criteria:

  * Recurrent disease
  * Stage IIIB with pleural or pericardial effusion
  * Stage IV disease
* Treated on protocol ECOG-2598

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-02-02 (Actual); Primary Completion 2006-07-02 (Actual); Study Completion 2006-07-02 (Actual)

PRIMARY OUTCOMES:
Correlation of HER-2 mutation with response, time to progression, and survival

CONTACTS AND LOCATIONS:
Overall Officials: David P. Carbone, MD, PhD, Study Chair — Vanderbilt-Ingram Cancer Center